CLINICAL TRIAL: NCT05279846
Title: A Multi-center, Double-blind, Randomized, Vehicle-controlled Study of Efficacy and Safety of Topical MOB015B in the Treatment of Mild to Moderate Distal Subungual Onychomycosis (DSO)
Brief Title: A Vehicle-controlled Study of Topical MOB015B in the Treatment of Distal Subungual Onychomycosis (DSO)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOB015B-33-21-001
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Onychomycosis
Keywords: Nail Fungus; Antifungal; Terbinafine; Distal Subungual Onychomycosis (DSO)
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MOB015B (Experimental): Applied at bedtime daily for 8 weeks and then reduced to once weekly for 40 weeks
  Interventions: Drug: MOB015B
- Control Arm (Placebo Comparator): Applied at bedtime daily for 8 weeks and then reduced to once weekly for 40 weeks
  Interventions: Drug: Vehicle (Placebo Comparator)

INTERVENTIONS:
Drug: MOB015B — Applied topically for 48 weeks
  Arms: MOB015B
Drug: Vehicle (Placebo Comparator) — Applied topically for 48 weeks
  Arms: Control Arm

SUMMARY:
This is a Phase 3 multicenter, double-blind study to evaluate the safety and efficacy of vehicle-controlled topical MOB015B in the treatment of Distal Subungual Onychomycosis (DSO)

DETAILED DESCRIPTION:
Distal subungual onychomycosis (DSO) is the most common form of Onychomycosis, in which fungi invade the underside of the nail plate. The infection may worsen, spread to other uninfected areas or infect other people. Without treatment the disease may have an impact on an individual's quality of life. MOB015B is a newly developed topical solution for the treatment of nail fungus (onychomycosis) containing the active antifungal ingredient terbinafine. All ingredients in MOB015B have a well-established use in approved pharmaceuticals for dermatological use. The purpose of this study is to evaluate the efficacy and safety of a new reduced dose treatment regimen of MOB015B whereby the investigational medicinal product (IMP) is applied daily for 8 weeks and then reduced to once weekly treatment for 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 12 to 75 years of age
2. Distal subungual onychomycosis of at least one of the great toenail(s) affecting 20% to 60% of the target great toenail (verified by a central blinded assessor before randomization)
3. Positive KOH microscopy and culture for dermatophytes in the target toenail
4. Ability of the great toenail to grow (e.g., subject reports cutting toenails at least monthly)
5. Signed written informed consent and assent (if applicable)

Exclusion Criteria:

1. Proximal subungual onychomycosis, superficial white onychomycosis, or significant dystrophy judged clinically by the blinded assessor or by the Investigator that may interfere with clinical evaluation of onychomycosis
2. Distal subungual onychomycosis where disease involvement has extended into the proximal portion of the target toenail and the unaffected proximal nail is less than 3 mm measured from proximal nail fold
3. Target toenail thickness more than 3 mm measured at the distal end
4. "Spike" of onychomycosis extending to eponychium of the target toenail
5. Presence of dermatophytoma (defined as thick masses of fungal hyphae and necrotic keratin) or severe onychorrhexis on the target toenail
6. Nail conditions other than DSO that are known to cause abnormal nail appearance, presence of melanonychia or subungual hematoma that could obscure visualization of nail clearing
7. Other microbial infections of the target toenail, for example, candida or mold infections without isolation of a dermatophyte
8. Previous target toenail surgery (within 6 months) with any residual disfigurement that will impact efficacy outcome or will not allow nail to grow normally, as judged by the Investigator
9. Topical treatment of the toenails with other antifungal medication within 6 weeks before Screening/Visit 1
10. History of failing oral therapy for onychomycosis within the past 3 years, or inability for nail to appear normal due to trauma, as judged by the Investigator
11. Systemic use of antifungal treatment within 6 months before Screening/Visit 1
12. Moderate to severe moccasin tinea pedis that require prolonged topical antifungal treatment or oral antifungal treatment should be excluded. Subjects with symptomatic interdigital tinea pedis or mild moccasin type tinea pedis will be screen failed. However, However, they will be allowed to enter the study after appropriate effective treatment and washout period as per Investigator judgment.
13. Signs of severe peripheral circulatory insufficiency as determined by significantly diminished/lack of pedal pulse on either foot
14. Subjects with a current or past history of psoriasis and/or lichen planus
15. Subjects with poorly controlled (or uncontrolled) diabetes mellitus as determined by HbA1c of > 8%
16. Known immunodeficiency, i.e., congenital immunodeficiency, acquired immunodeficiency, iatrogenic by immunosuppressive drugs like cytostatics or by radiation therapy or immunomodulatory medications (e.g., TNF inhibitors)
17. Participation in another clinical trial with an investigational drug or device during the previous 3 months before enrollment/baseline and for the duration of this study
18. Known allergy to any of the tested treatment products
19. Female subjects who are pregnant or breastfeeding; or intend to conceive a child during the duration of the study (52 weeks).
20. Subjects previously randomized to any study involving MOB015B treatment/exposure
21. History of, or current drug or alcohol abuse that would interfere with a subject's ability to participate in the study as determined by the Investigator
22. Psychiatric condition that might limit the participation in the study and/or that lead to the assumption that the subject's ability to completely understand the consequences of consent is missing
23. Close affiliation with the Investigator (e.g., a close relative) or persons working at the same study site, or subject who is an employee of the Sponsor/designee
24. Subjects who are institutionalized because of legal or regulatory order
25. Any diseases or circumstances in which the subject should not participate in the study in the opinion of the Investigator

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete cure of the target toenail | 52 Week
  Defined as negative fungal culture of dermatophytes, negative direct potassium hydroxide [KOH] microscopy and 0% clinical disease involvement
Incidence of adverse events (Safety) | 52 Week
  Safety as determined by the incidence of adverse events (AEs)

SECONDARY OUTCOMES:
Proportion of subjects with mycological cure of target toenail | 52 Week
  Defined as negative fungal culture of dermatophytes and negative direct KOH microscopy)
Proportion of subjects with treatment success of target toenail | 52 Week
  Defined as nails that are "completely clear" or "almost clear" of clinical diseases and negative mycology

CONTACTS AND LOCATIONS:
Locations (35):
- United States (33):
  - University of Alabama Hospital, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Center for Dermatology Clinical Research,Inc, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Center for Clinical Research, San Francisco, California
  - Colorado Medical Research Center, Denver, Colorado
  - Olympian Clinical Research, Clearwater, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Doctors Research Institute Corporation, South Miami, Florida
  - Podiatry 1st, O'Fallon, Illinois
  - The South Bend Clinic, LLC, South Bend, Indiana
  - DelRicht Research - Baton Rouge, Baton Rouge, Louisiana
  - IMA Clinical Research, Monroe, Louisiana
  - David Fivenson, MD, Dermatology, PLLC, Ann Arbor, Michigan
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Associated Skin Care Specs, New Brighton, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Hassman Research Institute, Berlin, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Weill Cornell Medicine Dermatology, New York, New York
  - Skin Search of Rochester, Rochester, New York
  - UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - Haber Dermatology, Inc., Beachwood, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Futuro Clinical Trials LLC, McAllen, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Houston Center for Clinical Research, Sugar Land, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (2):
  - Mediprobe Research, London, Ontario
  - Toronto Research Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No